CLINICAL TRIAL: NCT05541107
Title: Encochleated Oral Amphotericin for Cryptococcal Meningitis Trial 3
Acronym: EnACT3
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Matinas BioPharma Nanotechnologies, Inc. (Industry)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MB-70018; CTA 0217 (Other: Uganda National Drug Authority (NDA))
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Cryptococcal Meningitis
MeSH Terms: conditions — Meningitis, Cryptococcal | interventions — Amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MAT2203 Induction / MAT2203 Consolidation (Experimental): 2 days IV Amphotericin B (AMB) + flucytosine (5FC) followed by oral MAT2203 + 5FC for 12 days of induction therapy followed by MAT2203 +fluconazole for 4 weeks of consolidation therapy
  Interventions: Drug: MAT2203
- MAT2203 Induction / SOC Consolidation (Experimental): 2 days IV AMB + 5FC followed by oral MAT2203 + 5FC for 12 days of induction therapy followed by 4 weeks of standard of care consolidation therapy
  Interventions: Drug: MAT2203
- SOC Induction / SOC Consolidation (Active Comparator): Standard of care induction therapy (IV AMB + 5FC) followed by 4 weeks of standard of care consolidation therapy (fluconazole)
  Interventions: Drug: Amphotericin B

INTERVENTIONS:
Drug: MAT2203 — oral lipid nanocrystal amphotericin B
  Other Names: cAMB
  Arms: MAT2203 Induction / MAT2203 Consolidation; MAT2203 Induction / SOC Consolidation
Drug: Amphotericin B — Intravenous Amphotericin B
  Arms: SOC Induction / SOC Consolidation

SUMMARY:
This pivotal, confirmatory trial seeks to independently verify the results observed in the EnACT Phase II Stage 2 trial (MB-70007).

DETAILED DESCRIPTION:
Pivotal, prospective, randomized, open-label, non-inferiority trial to compare the efficacy and safety of step-down induction and consolidation therapy for the treatment of cryptococcal meningitis with oral MAT2203 plus flucytosine to standard of care therapy. Randomization will by 1:1:1 to one of two experimental arms or standard of care.

ELIGIBILITY:
Inclusion Criteria:

* CSF cryptococcal antigen (CrAg) positive meningitis
* Ability and willingness to provide informed consent
* Willing to receive protocol-specified lumbar punctures

Exclusion Criteria:

* Glasgow Coma Scale < 15 at time of consent
* Received >= 3 doses of amphotericin B within prior 30 days
* Inability to take enteral (oral or nasogastric) medicine
* Cannot or unlikely to attend regular clinic visits
* Receiving chemotherapy or corticosteroids
* Suspected paradoxical immune reconstitution inflammatory syndrome (IRIS)
* Pregnancy or breastfeeding
* Previous administration of MAT2203
* Any condition for which participation would not be in the best interest of the participant or that could limit protocol specified assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Survival | 2 weeks
  All-cause mortality

SECONDARY OUTCOMES:
Meningitis-free survival | 10 weeks
  Survival time without Cryptococcus culture-positive relapse of meningitis
Evidence of fungicidal activity | 2 weeks
  Rate of CSF Cryptococcus clearance (early fungicidal activity [EFA])
CSF culture sterility | 10 weeks
  cumulative incidence of CSF culture sterilization

CONTACTS AND LOCATIONS:
Overall Officials: David R Boulware, MD, Principal Investigator — University of Minnesota; David B Meya, MBChB, Principal Investigator — Infectious Diseases Institute

IPD SHARING:
Plan to Share IPD: No